CLINICAL TRIAL: NCT03672162
Title: Comparison of Effectiveness of Preoperative Gabapentin With Celecoxib in Reducing Acute Postoperative Pain in Abdominal Hysterectomy, A Randomized Double Blindcontrolled Trial
Brief Title: Preoperative Analgesia in Non-gynecological Cancerous Women Who Underwent Elective Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GabaCele
Record Dates: First submitted 2018-08-29; First posted 2018-09-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2018-08

CONDITIONS: Total Abdominal Hysterectomy ,Pain , Acute Postoperative,Gabapentin , Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gabapentin Group (Active Comparator): Subjects will receive Gabapentin 600 mg (two capsules of Gabapentin 300 mg) at two hours prior to surgery with clear water 30 ml and undergo elective total abdominal hysterectomy
  Interventions: Procedure: Total abdominal hysterectomy
- Celecoxib Group (Active Comparator): Subjects will receive Celecoxib 400 mg (two capsules of Celecoxib 200 mg) at two hours prior to surgery with clear water 30 ml and undergo elective total abdominal hysterectomy
  Interventions: Procedure: Total abdominal hysterectomy
- Placebo group (Placebo Comparator): Subjects will receive Placebo (two capsules of placebo) at two hours prior to surgery with clear water 30 ml and undergo elective total abdominal hysterectomy
  Interventions: Procedure: Total abdominal hysterectomy

INTERVENTIONS:
Procedure: Total abdominal hysterectomy — Each drug group undergo elective total abdominal hysterectomy with the same general anesthesia

SUMMARY:
Comparison of effectiveness of preoperative Gabapentin with Celecoxib in reducing acute postoperative pain in abdominal hysterectomy, A randomized double blind controlled trial

DETAILED DESCRIPTION:
Total abdominal hysterectomy (TAH) is the most common gynecological operation worldwide.Some studies noticed about overused of opioids in postoperative care , leaded to more adverse effect of opioids , slowly recovery , prolong length of hospitalized stay and consequently increase unnecessary cost of treatment.

ERAS guidelines has considered to use preoperative analgesics for reducing post-operative opioids consumption, including Gabapentin and Celecoxib.

Gabapentin and celecoxib widely used for treatment of pain and many studies have demonstrated the preoperative efficacy and safety of Gabapentin and Celecoxib in variety procedures involving hysterectomy.However, no definite conclusion of optimal dose and timing for preopearive uptake ,apart from no good evidences based supported preoperative Gabapentin or Celecoxib in hysterectomy in Thailand . In addition, the protocol for preoperative analgesics in hysterectomy, has not been performed in the investigator's center.

Therefore the aim of this study is to assess and compare the efficacy and safety of preoperative Gabapentin and Celecoxib to reduce acute postoperative pain in non-gynecological cancerous woman undergoing total abdominal hysterectomy

ELIGIBILITY:
Inclusion Criteria:

* Women ranging age between 18-65 years and having non-gynecological cancerous women who undergoing elective total abdominal hysterectomy
* Women who has ASA physical status I-II
* Women who agrees to participate in this study

Exclusion Criteria:

* Women who pregnancy
* Women who have abnormal kidney function test (Cr > 1.5 )
* Women who have abnormal liver function test
* Women with history or present of thrombosis such as myocardial infarction, ischemic stroke, deep venous thrombosis or pulmonic embolism
* Women with history of gastrointestinal bleeding -Women with history of gastrointestinal bleeding -Women with history of gastrointestinal bleeding
* Women who take the antiplatelet or anticoagulant medications
* Women with history of allergy to Gabapentin ,Celecoxib and Sulfa
* Women who have used or known Gabapentin or Celecoxib before
* Women who have chronic alcoholism
* Women who underwent previous surgery
* Women who undergo extended low midline incision
* Women who undergo lysis adhesion
* Women who undergo further operations except salpingo-oophorectomy
* Women who cannot evaluated pain score

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Subjective pain at 24 hours post operation: numeric analog scale | During acute post operation peroid as 24 hours post operation
  Assessment of subjective pain score post operation at 24 hours (at first visit at inpatient ward , 4,5,8,12 and 24 hours after surgery ),by using a numeric analog pain scale from .Score 0-10 .When Score is higher than 5 score ,the pateint will gain the analgesia as opioid

SECONDARY OUTCOMES:
Adverse effects of Gabepentin and Celecoxib at 24 hours post operation | During acute post operation peroid as 24 hours post operation
  Will assess for known symptoms of Gabapentin post operation 24 hours (at first visit at inpatient ward , 4,5,8,12 and 24 hours after surgery ).We will survey subjects regarding their experience of the following symptoms : nausea and vomiting ,dizziness, drowsiness ,allergic reaction ,chest pain ,and gastrointestinal bleeding .
First opioid rescue dose at 24 hours post operation | During acute post operation peroid as 24 hours post operation
  First time of reciving the opioid after surgery in 24 hours
Opioid consumption at 24 hours post operation (at first visit at inpatient ward , 4,5,8,12 and 24 hours after surgery ) | During acute post operation peroid as 24 hours post operation
  Total dose of opioid consumtion in 24 hours after surgery
Subjective pain at the time of discharge: numeric analog pain scale | Date of discharge ,not longer than 7 days after admit
  Assessment of subjective pain score at the time of discharge ,will use a numeric analog scale from 0-10 .
Length of hospitalization stay | Date from of admit to date of discharge,not longer than 7 days after admit
  measure days of hospitalization since date of admit to date of discharge in this visitting

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided